CLINICAL TRIAL: NCT04076605
Title: Bleeding in Hospitalized Patients With Liver Disease Undergoing Invasive Procedures
Acronym: PROC-BLeeD
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Nicolas Intagliata, MD, Associate Professor, Gastroenterology, University of Virginia
Other Study IDs: 21671
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Bleeding; Procedural Complication; Cirrhosis, Liver; Coagulation Disorder, Blood
Keywords: Decompensated; Liver; Coagulopathy; ACLF
MeSH Terms: conditions — Hemorrhage; Liver Cirrhosis; Blood Coagulation Disorders; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with cirrhosis are frequently hospitalized and often undergo procedures. Knowledge surrounding bleeding risk is sparse and practice patterns vary across centers in regards to bleeding prophylaxis. The goal of this study to is to obtain more knowledge regarding risk factors for procedural related bleeding in patients with cirrhosis and to develop a predictive model to risk stratify patients before undergoing procedures. Through collaboration from centers across the world this study should provide information on prevalence of bleeding and variation in practice patterns for prophylaxis.

DETAILED DESCRIPTION:
Hospitalized patients with cirrhosis who undergo 1 or more non-surgical procedure will be enrolled. The investigators will collect multiple clinical characteristics from the medical record and follow the patients prospectively over the hospitalization and/or until 28 days to determine if clinical events have occurred including bleeding, thrombosis, re-hospitalization and death. Characteristics of the hospitalization will be recorded including presence of acute decompensation and acute on chronic liver failure (ACLF). Procedure type will be recorded including coagulation laboratory data before and after each procedure. All bleeding events will be recorded and characteristics surrounding each bleed will be recorded. Bleeding will be defined according to International Thrombosis and Haemostasis (ISTH) definitions of major bleed and clinically relevant non-major bleed. REDCap (https://www.project-redcap.org) will be used to collect and centralize data maintained at the University of Virginia. Characteristics of each hospitalization will be recorded accordingly and patients will be followed for 28 days for outcome and mortality information. Each participating center will obtain local Institutional Review Board (IRB) approval to participate and enter data directly into REDCap. After center IRB approval is obtained, centers will consecutively enrolling patients on a rolling basis. Data will be collected from enrollment until death, transplant, discharge and/or 28 days on each individual enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with cirrhosis admitted to a hospital ward or ICU for greater than 24 hours.
* Patient must undergo 1 or more invasive non-surgical procedures at admission or during the hospitalization.

Exclusion Criteria:

* Age < 18 years old
* Prisoner
* Pregnant
* Unable to provide consent
* Previously enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cirrhosis admitted to the hospital are evaluated and then consented to participate in the study (see Inclusion/Exclusion). Patients with cirrhosis admitted to the general ward or intensive care unit may be enrolled.
  The investigators will collect multiple clinical characteristics from the medical record and follow the patients over the hospitalization and/or until 28 days to determine if clinical events have occurred including bleeding, thrombosis, re-hospitalization and death.
Sampling Method: Non-Probability Sample
Enrollment: 1182 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of procedural-related bleeding events in patients with cirrhosis | Each patient enrolled will be followed for 28 days
  During each hospitalization every procedure will be recorded and details surrounding each bleeding event related to a procedure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas M Intagliata, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States